CLINICAL TRIAL: NCT07192913
Title: Investigating the Impact of Transcranial Magnetic Stimulation (TMS) on Amyloid and Tau Clearance Via Glymphatic Function in Prodromal Alzheimer's Disease
Brief Title: Glymphatic Function TMS Study
Acronym: GF-TMS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Ying-hui Chou, Principle Investigator, University of Arizona
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 25103278; 022713-00001 (Other Grant/Funding Number: Arizona Alzheimer's Consortium)
Record Dates: First submitted 2025-09-12; First posted 2025-09-25 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active (TBS) - Sham (TBS) (Experimental): Block 1: Active TBS Block 2: Sham TBS
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham (TBS) - Active (TBS) (Experimental): Block 1: Sham TBS Block 2: Active TBS
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — TMS is a non-invasive brain stimulation technique. The primary aim of the study will be to verify the deliverability of the TMS effect on the hippocampus and determine which stimulation protocol is more beneficial to each participant.
  Device: Transcranial Magnetic Stimulation (Sham)
  TMS is a non-invasive brain stimulation technique. The primary aim of the study will be to verify the deliverability of the TMS effect on the hippocampus and determine which stimulation protocol is more beneficial to each participant. For sham, the side of the coil that does not deliver pulses will be used.

SUMMARY:
The purpose of this study is to use transcranial magnetic stimulation (TMS) in older adults to impact the glymphatic system. The glymphatic system is a brain-wide clearance pathway that plays a crucial role in removing dysfunctional proteins in Alzheimer's disease. This project aims to investigate if TMS can help glymphatic function and reduce levels of these proteins in those with mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

Individuals with mild cognitive impairment (MCI Group)

Inclusion Criteria:

* Age 18-85 years
* MCI subjective criteria: self- or informant-reported cognitive complaint
* Objective cognitive impairment supported by one of the following measures of general cognitive function: (a) classified as MCI via the NACC-UDS 3.0 neuropsychological battery using the typical neuropsychological criteria for MCI diagnosis (1 score on any test at least1.5 SD below the mean); or (b) classified as MCI via the NACC-UDS 3.0 neuropsychological battery using the Jak/Bondi neuropsychological criteria for MCI diagnosis(2 scores at least 1 SD below the mean in one domain, or 3 scores at least 1SD below the mean across domains)
* Right-handed
* English speaking
* Able to attend daily intervention and outcome measurements for ~15 days over a 6 month period.
* Not enrolled in another interventional study within 6 months prior to beginning this study

Exclusion Criteria:

* Contraindications to transcranial magnetic stimulation (TMS) or magnetic resonance imaging (MRI)
* Reported sudden or steep decline of cognitive performance
* Telephone Interview for cognitive impairment (TICS) score
* Other neurological disorders (e.g., stroke, head injuries, or multiple sclerosis)
* Psychiatric disorder (except stable late-life depression due to its high prevalence in MCI individuals)
* Current cancer treatment or other comorbid/unstable medical conditions that might independently affect cognitive function

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
NIH Toolbox | Day 1(baseline for block 1), Day 14(post block 1), Day 70 (Baseline block 2), Day 84 (post block 2)
  The NIH Toolbox Cognition Battery, recommended for ages 7+, consists of tests of multiple constructs. It yields individual test scores and the following summary scores: Total Cognition Composite, Fluid Composite (includes Dimensional Change Card Sort, Flanker Inhibitory Control and Attention, Picture Sequence Memory (Form A), List Sorting Working Memory, and Pattern Comparison tests), and Crystallized Composite (includes Picture Vocabulary and Oral Reading Recognition tests).

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Hui Chou, Sc.D., Principal Investigator — University of Arizona

IPD SHARING:
Plan to Share IPD: No
N/A Will not be sharing data